CLINICAL TRIAL: NCT00741312
Title: Influence of Physical Exercise on Endothelial Function in Pregnant Women: Randomized Clinical Trial
Brief Title: Influence of Physical Exercise on Endothelial Function in Pregnant Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Ana Cecilia Aguilar de Plata, Universidad del Valle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 182-07
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Pregnancy; Preeclampsia; Exercise
Keywords: pregnancy; preeclampsia; exercise
MeSH Terms: conditions — Pre-Eclampsia; Motor Activity | interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental)
  Interventions: Behavioral: Regular aerobic physical exercise
- II (Active Comparator)
  Interventions: Behavioral: Activities of daily living

INTERVENTIONS:
Behavioral: Regular aerobic physical exercise — Walking (10 minutes), aerobic exercise (30 minutes), stretching (10 minutes) and relaxation exercise (10 minutes). Exercise will be performed at three sessions per week. All sessions will be supervised by a physical therapist and a physical educator.
  The exercise-program follows the ACOG and ACSM exercise prescription. Aerobic activities will be performed at moderate intensity (60-70% of maximal heart rate) measured by the 6-20 Borg's rating scale. Each session starts with a 5 minutes of warm up, followed by 30 minutes of aerobic activity, including 5 minutes cool down. This is followed by 15 minutes of circuit strength training of the upper limbs, lower limbs, and deep abdominal stabilization muscles. The last 5 minutes consists of stretching and relaxation exercises.
  Arms: I
Behavioral: Activities of daily living — Basic activities of daily living (bathing, dressing, eating, walking) without counseling by a physical therapist.
  Arms: II

SUMMARY:
The purpose of this study is to determine the effect of regular aerobic exercise on endothelial function in pregnancy.

DETAILED DESCRIPTION:
Preeclampsia is a common maternal disease that complicates 5% to 10% of pregnancies and remains as the major cause of maternal and neonatal mortality, especially in developing countries. Cost-effective interventions aimed to prevent the development of preeclampsia are urgently needed. Ethiopathogenesis of preeclampsia involves multiple mechanisms as oxidative stress, endothelial dysfunction, infections, maternal constitutional factors, and others. Regular aerobic exercise recovers endothelial function, decreases oxidative stress and improves maternal constitutional factors.

The purpose of this Controlled Clinical Trial is to determine the effect of regular aerobic exercise on endothelium-dependent brachial artery flow-mediated dilatation. Furthermore, the effect of exercise on biomarkers on vascular function and perinatal outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who have not participated in a structured exercise program, including significant amounts of walking for the past four months are eligible for the trial.
* Live foetus at the routine ultrasound scan and a normal pregnancy.
* Gestational age 16 to 20 weeks
* Written informed consent will be obtained from each woman prior to the inclusion in the study.

Exclusion Criteria:

* History of high blood pressure
* Chronic medical illnesses (cancer, renal, endocrinologic, psychiatric, neurologic, infectious and cardiovascular diseases)
* Persistent bleeding after week 12 of gestation
* Poorly controlled thyroid disease
* Placenta praevia, incompetent cervix, polyhydramnios, oligohydramnios
* History of miscarriage in the last twelve months
* Diseases that could interfere with participation (following recommendations from ACSM 2000, ACOG 2003).

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | Baseline, 8 weeks, 16 weeks

SECONDARY OUTCOMES:
high sensitivity C-Reactive Protein | Baseline, 16 weeks
Nitrates, Nitrites and cyclic GMP | Baseline, 16 weeks
Blood lipid profile | Baseline, 16 weeks
Anthropometric indicators | Baseline, 8 weeks, 16 weeks
Functional capacity (VO2 Max) | Baseline, 8 weeks, 16 weeks
Maternal and neonatal outcomes | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Plata, MSc, Principal Investigator — Universidad del Valle; Adalberto Sanchez, PhD, Principal Investigator — Universidad del Valle
Locations (1):
- Centro de Salud Cañaveralejo, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Pinzon DC, Zamora K, Martinez JH, Florez-Lopez ME, de Plata AC, Mosquera M, Ramirez-Velez R. Type of delivery and gestational age is not affected by pregnant Latin-American women engaging in vigorous exercise: a secondary analysis of data from a controlled randomized trial. Rev Salud Publica (Bogota). 2012 Oct;14(5):731-43. PMID 24652353
- [Derived] Montoya Arizabaleta AV, Orozco Buitrago L, Aguilar de Plata AC, Mosquera Escudero M, Ramirez-Velez R. Aerobic exercise during pregnancy improves health-related quality of life: a randomised trial. J Physiother. 2010;56(4):253-8. doi: 10.1016/s1836-9553(10)70008-4. PMID 21091415
- [Derived] Ramirez-Velez R, Aguilar AC, Mosquera M, Garcia RG, Reyes LM, Lopez-Jaramillo P. Clinical trial to assess the effect of physical exercise on endothelial function and insulin resistance in pregnant women. Trials. 2009 Nov 17;10:104. doi: 10.1186/1745-6215-10-104. PMID 19919718